CLINICAL TRIAL: NCT01758068
Title: Effect of Topical Oil Application on Trans-Epidermal Water Loss in Preterm Infants - A Randomized Clinical Trail
Brief Title: Effect of Twice Daily Application of Coconut Oil in Reducing Water Loss From Skin of Premature Babies in First Week of Life
Acronym: TEWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Collaborators: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Professor, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AIIMS/06/TEWL
Record Dates: First submitted 2012-12-23; First posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Trans Epidermal Water Loss
Keywords: Preterms; Coconut Oil application; Trans epidermal water loss; Weight gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coconut Oil Application (Experimental): The oil (coconut oil) was applied by the trained nurse to the entire body surface of infant except the face two times a day started as early as possible Four ml of coconut oil was applied using both hands of the caregiver in four strokes starting from the level of clavicles over the chest and abdomen till the groin, from the front of thighs, knee, leg and upto the sole, from above the shoulders over the arm and forearm till the palm continuing medially over the forearm and arm till the axilla and the final stroke was used for the back reaching over the back of the thighs till the heel. Just prior to the first application, and thereafter prior to the subsequent applications the TEWL was recorded using the portable closed chamber evaporimeter. The oil application was continued twice daily (every 12 hrs at the same time as the hour of birth e.g. 11 am and 11pm) till the completion of the seventh day (168 hrs of life)..
  Interventions: Procedure: Coconut Oil Application
- No Oil Application (No Intervention): Babies in this group were not subjected to oil application. TEWL measurement was recorded every 12 hrs for the first week of life, at the same time as the hour of birth.

INTERVENTIONS:
Procedure: Coconut Oil Application — Coconut oil - 4 ml
  Arms: Coconut Oil Application

SUMMARY:
The skin of newborn infants is immature and ineffective as a barrier. Preterm skin exhibits even more vulnerability to the environment due to poor self regulatory heat mechanisms, paucity of fatty tissue and its thinness. Most preterm babies lose up to 13% of their weight as water loss from their skin during the first week of life. Many strategies have been utilized by neonatologists to decrease this water loss. Edible coconut oil application on the skin acts as a non permeable barrier and can help in achieving this. Hence the investigators decided to undertake this study to objectively assess the reduction in water loss from skin after oil application.

ELIGIBILITY:
Inclusion Criteria:

All preterm babies born at the study center with birth weight < 1500g were eligible for inclusion in the study.

Exclusion Criteria:

1. Babies with birth weight less than 750 gms at birth
2. Babies with major congenital malformations.
3. Babies with severe asphyxia, hydrops and shock.
4. Babies with congenital diseases of skin associated with skin breach or denudation of skin precluding oil application
5. Babies with preexisting skin infection such as multiple furuncles (2 or more skin areas - each limb, head, chest, abdomen and back are the individual areas that will be taken as one area)

Ages: 12 Hours to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2005-11; Primary Completion 2006-09 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Trans Epidermal Water Loss(TEWL) | first 7 days of life
  TEWL was measured using evaporimeter(Vapometer, Delfin Technologies limited, Kuopio, Finland) at 12 hours of age and thereafter every 12 hours till first 7 days of life

SECONDARY OUTCOMES:
Weight | first 7 days of life and 40 weeks postmenstrual age
  The weight of the neonate was recorded at birth and daily during the first week of life. The weight in grams and weight gain in grams/kilogram/day was measured at 40 weeks post conceptional age.
Skin condition Score | at day 7 of life
  Skin Condition Score was measured using 'Lane and Drost' Score.This score has 9 scores from 1 to 9, 1 depicting the best skin state and 9 the worst with erythema, blistering & oozing over the entire area.
Skin colonization pattern | at day 7 of life
  The skin swab cultures were sent after 1week of life to assess for skin colonization

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, MD, DM, Principal Investigator — All India Institute of Medical Sciences

REFERENCES:
- [Derived] Nangia S, Paul VK, Deorari AK, Sreenivas V, Agarwal R, Chawla D. Topical Oil Application and Trans-Epidermal Water Loss in Preterm Very Low Birth Weight Infants-A Randomized Trial. J Trop Pediatr. 2015 Dec;61(6):414-20. doi: 10.1093/tropej/fmv049. Epub 2015 Sep 3. PMID 26338490